CLINICAL TRIAL: NCT02753491
Title: The Effect of Motivational Short Interview Model in Type 2 Diabetic Paitent in Primary Care in TURKEY
Brief Title: The Effect of Motivational Short Interview Model in Type 2 Diabetic Patient in Primary Care in TURKEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2015.218
Record Dates: First submitted 2016-04-24; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Lifestyle-related Condition
Keywords: short interview, diabetes, lifestyle changes, primary care
MeSH Terms: conditions — Mental Disorders; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): In intervention group, three or four motivational short interview made with every participants.
  Interventions: Behavioral: Motivational short interview
- Control (No Intervention): non intervention group,

INTERVENTIONS:
Behavioral: Motivational short interview — New designed motivational short interview model
  Arms: Intervention

SUMMARY:
This study designed for primary care practionars for chronic care in primary care. A new model of motivational short interview used for intervention. The aim of this study is to develop diet and exercise regimens in type 2 diabetic patients.

DETAILED DESCRIPTION:
This is a randomized controlled trial. The pedometer for one week has given to and filling one day food intake form asked from all participants. The weights and the heights of the participants were measured and the Beck depression scale for primary care, the modify Moresby scale, the EQ5D, the MDDQ and the motivation scale filled face to face with all participants. In intervention group the steps of the motivational short interview model were; increase patient awareness about his/her type 2 diabetes and its difficulties, then discuss alternative solutions for the problems the participant has and making decisions for action, and the third and fourth interview includes new alternative solutions for new difficulties if there is and promotion of self efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Being type 2 diabetic unless for one year
* No drug changes for last three months
* HbA1c levels between 7-10%
* BMI >25 kg/m2
* At least %80 compliance with medical treatment
* no depression

Exclusion Criteria:

* Getting >7 point from beck depression scale for primary care
* Using anti depressed treatment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
increasing pedometer levels +1300 step | 3 months
  increasing one week pedometer mean + 1300 step using short interview model
decreasing 300 cal daily food intake | 3 months
  decreasing 300 cal daily food intake using short interview model

SECONDARY OUTCOMES:
increasing short EPAQ category to 2 from 1. | 3 months
loosing weight | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet AKMAN, Asis. Prof., Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No